CLINICAL TRIAL: NCT00418210
Title: A Multicentre Feasibility Study of Accelerated Partial Breast Irradiation Using Three-dimensional Conformal Radiation Therapy for Early Breast Cancer.
Brief Title: Accelerated Partial Breast Irradiation for Early Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 06.02; ACTRN12607000238471 (Registry Identifier: ANZ CTR)
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer
Keywords: Accelerated Partial Breast Irradiation; Conformal Radiation Therapy; Feasibility; Early breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Conformal; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Accelerated partial breast irradiation (Experimental): Accelerated partial breast irradiation (APBI) to region of tumour bed using 3D conformal radiation therapy (3D CRT)
  Interventions: Radiation: Accelerated partial breast irradiation (APBI) to region of tumour bed using 3D conformal radiation therapy (3D CRT)

INTERVENTIONS:
Radiation: Accelerated partial breast irradiation (APBI) to region of tumour bed using 3D conformal radiation therapy (3D CRT) — Accelerated partial breast irradiation (APBI) to region of tumour bed using 3D conformal radiation therapy (3D CRT; 38.5 Gy in 3.85 Gy fractions bi-daily over 5 consecutive working days
  Other Names: Radiation

SUMMARY:
Hypothesis:

In selected women with node-negative invasive breast cancer treated with breast conserving surgery, postoperative accelerated partial breast irradiation (APBI) limited to the region of the tumour bed delivered by 3-dimensional conformal radiation therapy (3D CRT) is technically feasible and reproducible with acceptable treatment toxicity, cosmetic outcome, and local control rate in a multicentre trial.

DETAILED DESCRIPTION:
This is a TROG multicentre feasibility study of APBI using 3D CRT in selected women with node-negative breast cancer treated by breast conserving surgery with negative margins.

This is a one-arm feasibility study in which the primary endpoint is the feasibility rate for APBI using 3D CRT. This is defined as the proportion of eligible patients treated without a major protocol deviation. Secondary endpoints include radiation toxicity, cosmetic outcome, quality of life, time to ipsilateral breast recurrence, disease-free survival, and overall survival.

Primary objectives: To evaluate the technical feasibility and reproducibility of APBI limited to the region of the tumour bed using 3D CRT following breast conserving surgery.

Secondary objectives:

* To assess the acute and long term toxicity of APBI using 3D CRT.
* To examine the cosmetic outcome of women with breast cancer treated by breast conserving surgery and APBI using 3D CRT.
* To determine the time to ipsilateral breast recurrence, disease free survival and overall survival of women with node-negative breast cancer completely resected by breast conserving surgery followed by APBI using 3D CRT.
* To assess the quality of life of women with node-negative breast cancer treated by breast conserving surgery and APBI using 3D CRT.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all of the following criteria for admission to study:

* Women aged >= 50 years.
* Histologically confirmed diagnosis of invasive breast carcinoma of non-lobular histology.
* Bilateral mammograms performed within 6 months prior to registration.
* Treated with breast conserving surgery (primary excision or re-excision) with negative radial resection margins of >= 2 mm* for both the invasive and if present, associated intraductal tumour.

  *Patients with superficial or deep resection margin of < 2 mm are eligible if surgery has removed all of the intervening breast tissue from the subcutaneous tissue to the pectoralis fascia.
* Unifocal tumour measuring ≤ 20 mm in maximum microscopic dimension.
* Negative nodal status determined by sentinel node biopsy, axillary dissection, or for women > 70 years of age, clinical examination.
* No evidence of distant metastasis.
* Assessed by surgeon and radiation oncologist to be suitable for breast conserving therapy.
* Ability to tolerate protocol therapy.
* Protocol therapy must commence no later than 12 weeks from the last surgical procedure or 8 weeks from the last dose of chemotherapy.
* Availability for long-term follow-up.
* Women of child-bearing potential must use adequate contraception during RT.
* Written informed consent.

Exclusion Criteria:

Patients who fulfill any of the following criteria are not eligible for admission to study:

* Multifocal or multicentric tumours.
* Clinical or pathologic evidence of any of the following tumour features: extension to chest wall (excluding pectoralis muscle); oedema (including peau d'orange) or ulceration of skin; satellite skin nodules confined to the same breast; and inflammatory carcinoma.
* Presence of extensive intraductal component (ductal carcinoma in situ occupying > 25% of the primary invasive tumour and present adjacent to the primary tumour).
* Node-positive breast cancer determined by sentinel node biopsy, axillary dissection, or in women > 70 years of age, clinical examination.
* Inability to localise surgical cavity on CT scans with no evidence of a surgical cavity, seroma or surgical clips delineating the tumour bed.
* Treatment target volume estimated to occupy > 25% of the ipsilateral whole breast volume.
* Synchronous or metachronous bilateral invasive or intraductal breast cancer.
* Locally recurrent breast cancer.
* Ipsilateral breast implant.
* Serious non-malignant disease that precludes definitive surgical or radiation treatment (e.g. scleroderma, systemic lupus erythematosus, cardiovascular/pulmonary/renal disease).
* Previous or concomitant malignancies except non-melanoma skin cancer, carcinoma in situ of the cervix, and invasive carcinoma of the colon, thyroid, cervix, or endometrium treated five years prior to study entry.
* Women who are pregnant or lactating.
* Psychiatric or addictive disorders that preclude obtaining informed consent or adherence to protocol

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-08; Primary Completion 2018-06 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Feasibility rate of APBI using 3D conformal radiation therapy | First analysis will occur 6 months after accrual of all patients (approximately 1.5 years after start of trial)

SECONDARY OUTCOMES:
Radiation toxicity | First analysis will occur 6 months after accrual of all patients (approximately 1.5 years after start of trial). A final analysis will occur when all patients have been followed up for 5 years.
Cosmetic outcome | First analysis will occur 5 years after accrual of all patients (approximately 6 years after start of trial)
Quality of life | First analysis will occur 5 years after accrual of all patients (approximately 6 years after start of trial). A final analysis will occur when all patients have been followed up for 5 years.
Time to ipsilateral breast recurrence | First analysis will occur 5 years after accrual of all patients (approximately 6 years after start of trial). A final analysis will occur when all patients have been followed up for 5 years.
Disease free survival | First analysis will occur 5 years after accrual of all patients (approximately 6 years after start of trial). A final analysis will occur when all patients have been followed up for 5 years.
Overall survival | A final analysis will occur when all patients have been followed up for 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Boon Chua, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (7):
- Australia (5):
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Wooloongabba, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- New Zealand (2):
  - Auckland Hospital, Auckland
  - Waikato Hospital, Hamilton

REFERENCES:
- [Background] Kron T, Willis D, Miller J, Hubbard P, Oliver M, Chua B. A spreadsheet to determine the volume ratio for target and breast in partial breast irradiation. Australas Phys Eng Sci Med. 2009 Jun;32(2):98-104. doi: 10.1007/BF03178635. PMID 19623861
- [Result] Kron T, Willis D, Bignell F, Martland J, Donnell S, May S, Chua BH. Centre credentialing for Trans Tasman Radiation Oncology Group trial 06.02: multicentre feasibility study of accelerated partial breast irradiation. J Med Imaging Radiat Oncol. 2009 Aug;53(4):412-8. doi: 10.1111/j.1754-9485.2009.02097.x. PMID 19695049
- [Derived] Kron T, Willis D, Link E, Lehman M, Campbell G, O'Brien P, Chua B. Can we predict plan quality for external beam partial breast irradiation: results of a multicenter feasibility study (Trans Tasman Radiation Oncology Group Study 06.02). Int J Radiat Oncol Biol Phys. 2013 Nov 15;87(4):817-24. doi: 10.1016/j.ijrobp.2013.07.036. Epub 2013 Sep 21. PMID 24064318
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au